CLINICAL TRIAL: NCT06455176
Title: Delayed Secondary Reconstruction of Alveolar Clefts Using Autogenous Symphyseal Particulate Bone Versus Iliac Cancellous Bone: A Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Shawky, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo uni research
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Bone Facial Bone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symphyseal bone group (Active Comparator)
  Interventions: Procedure: alveolar cleft Grafting from the symphysis
- iliac cancellous bone group (Active Comparator)
  Interventions: Procedure: alveolar cleft Grafting from the iliac cancellous bone

INTERVENTIONS:
Procedure: alveolar cleft Grafting from the symphysis — grafting using particulate bone from the symphysis
  Arms: Symphyseal bone group
Procedure: alveolar cleft Grafting from the iliac cancellous bone — grafting using iliac cancellous bone
  Arms: iliac cancellous bone group

SUMMARY:
Patients with alveolar clefts whose ages are after 12 years (after eruption of all permanent dentition) were recruited and treated either by particulate bone grafting from the symphysis or from the anterior iliac crest

ELIGIBILITY:
Inclusion Criteria:

* cleft alveolus patients of both genders after eruption of all permanent dentition

Exclusion Criteria:

* previous failed repairs of alveolar clefts and bone metabolic diseases

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
bone volume in the reconstructed cleft site | six months

IPD SHARING:
Plan to Share IPD: Undecided